CLINICAL TRIAL: NCT02961504
Title: Placebo-Controlled, Double-Blind, Phase 2/3 Efficacy and Safety Trial of HLCM051 (MultiStem®) in Patients With Ischemic Stroke
Brief Title: Treatment Evaluation of Acute Stroke for Using in Regenerative Cell Elements
Acronym: TREASURE
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Healios K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B01-03
Record Dates: First submitted 2016-11-07; First posted 2016-11-11 (Estimated); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HLCM051 (MultiStem) (Experimental): single dose of 1.2 billion HLCM051 cells
  Interventions: Biological: HLCM051
- Placebo (Placebo Comparator): a single dose of placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: HLCM051 — Within 18 to 36 hours after the onset of ischemic stroke, subjects will receive a single dose of 1.2 billion HLCM051 cells to be intravenously administered
  Arms: HLCM051 (MultiStem)
Biological: Placebo — Within 18 to 36 hours after the onset of ischemic stroke, subjects will receive a single dose of placebo to be intravenously administered
  Arms: Placebo

SUMMARY:
The primary objectives of this study is to evaluate the efficacy of HLCM051 on functional outcome in subjects with acute ischemic stroke and to evaluate the safety of HLCM051 in subjects with acute ischemic stroke.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, multicenter, phase 2/3 trial to evaluate the efficacy and safety of intravenous administration of HLCM051 compared with placebo in subjects with acute ischemic stroke (within 36 hours of onset). Japanese subjects who developed a subcortical ischemic stroke and are eligible to participate in the trial will be evaluated.

Approximately 220 subjects will be randomized in a 1:1 ratio (HLCM051 group [n=110] or placebo group [n=110]) to receive a single infusion of HLCM051 or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male or female patients 20 years of age or older;
* Clinical diagnosis of cerebral cortical ischemic stroke;
* Occurrence of an ischemic stroke with clear motor or speech deficit documented by National Institutes of Health Stroke Scale (NIHSS) score of 8 to 20 (at the baseline assessment) that did not change by ≥4 points from the screening to the baseline assessment;
* Onset of ischemic stroke must have occurred within 18 to 36 hours prior to the start of administration of the investigational product;
* Confirmation of hemispheric cortical infarct with brain magnetic resonance imaging (MRI) including diffusion-weighted imaging with b-value of 1,000 demonstrating an acute lesion measuring ≥ 2.0 cm of longest diameter;
* A modified Rankin Scale (mRS) of 0 or 1, by either self-report or family report, prior to the onset of ischemic stroke;
* Female patients who meet either:

  * Not pregnant, not breastfeeding/ interrupting breastfeeding, and not planning on becoming pregnant during the trial;
  * Not of childbearing potential, defined as one who has been postmenopausal for at least 1 year, or has been surgically sterilized, or has had a hysterectomy at least 3 months prior to the start of this trial; or
  * If of childbearing potential, one who has agreed to follow investigator's advice and use an effective contraceptive method up to the end of the trial. Effective contraceptive methods include contraceptive methods used consistently and correctly (oral contraceptives, intrauterine devices, diaphragm, or male or female condoms), abstinence, and a sterile sexual partner;
* Male patients with female partners of childbearing potential must agree to follow investigator's advice and use adequate contraceptive methods (a combination of a condom and another form of contraception) up to the end of the trial if engaging in sexual intercourse;
* Patients or legal representatives must freely sign the informed consent form after the nature of the trial and the disclosure of his/her data have been explained;
* Willing and able to comply with all aspects of the treatment and testing schedule; and
* Willing and able to return to the trial site for the post-treatment evaluations.

Exclusion Criteria:

* Presence of a lacunar, a lesion of ≤ 2.0 cm of longest diameter, or a brainstem infarct on MRI as the etiology of symptoms of ischemic stroke;
* Reduced level of consciousness (score of 3 for item 1a of NIHSS);
* Occurrence of a hemorrhagic transformation as evidenced by computerized tomography (CT) or brain MRI scan that is clinically significant in the opinion of the investigator;
* Ipsilateral focal neurological deficits from prior lesions in the brain that would complicate evaluation;
* Experienced seizures since the onset of ischemic stroke;
* History of a neurological event such as stroke or clinically significant head trauma within 6 months prior to the start of screening;
* Patients who both received tPA treatment and underwent mechanical reperfusion (patients are eligible for the trial if they had only one of them, tPA treatment or mechanical reperfusion);
* Uncontrolled hypertension, defined as persistent systolic blood pressure >220 mmHg or diastolic blood pressure >120 mmHg, despite antihypertensive therapy;
* Blood glucose level <50 mg/dL or >350 mg/dL at baseline;
* Patients who have a significant comorbid medical condition(s), including, but not limited to:

  * Severe kidney disease requiring hemodialysis or peritoneal dialysis;
  * Advanced liver disease such as hepatitis or liver cirrhosis;
  * Severe congestive heart failure or history of ejection fraction <30%;
  * Severe lung disease requiring home oxygen; or
  * Active unstable angina requiring daily treatment with nitrates or other medications;
* Known human immunodeficiency virus infection, ongoing systemic infection, severe local infection or who are immunocompromised;
* Alzheimer's disease or other dementias, Parkinson's disease, or any other neurological disorder that in the opinion of the trial doctor would affect their ability to participate in the trial or confound study assessments;
* History of malignant tumor(s) within 2 years of the onset of ischemic stroke, with the exception of adequately treated basal or squamous cell carcinoma of the skin;
* Contraindication for MRI such as implanted pacemakers or other metallic prosthesis incompatible with MRI, body weight, or claustrophobia;
* Thrombocytopenia (platelet count <100,000/mm3) or heparin-induced thrombocytopenia;
* Known allergy to human tissue or bovine or porcine products, or religious objections to biological products;
* Prior participation in another clinical trial involving investigational pharmacological agents or devices within 30 days prior to providing consent to receive the investigational product, or participation in investigational pharmacological agents, devices, or rehabilitation stroke recovery program is planned during the trial;
* Other serious medical or psychiatric illness that is not adequately controlled and, in the investigator's opinion, would not permit the subject to be managed according to the protocol;
* Previous surgical removal of the spleen;
* Major fluctuation in neurological status since the onset of ischemic stroke indicating progression or expansion of ischemic stroke, or possible transient ischemic attack;
* Plan to have a neurovascular procedure (e.g., carotid endarterectomy, stent placement, etc.) within the first year following ischemic stroke; or
* Abnormal laboratory test results which investigators consider clinically significant and inappropriate for the trial.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2017-11-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects with an excellent outcome defined by the functional assessments | Day 90
  <Excellent outcome> is defined as mRS score of ≤1 (scale, 0 to 6), NIHSS score of ≤1 (scale, 0 to 42), and BI score of ≥95 (scale, 0 to 100).
Comparison between the HLCM051 and the placebo groups in key adverse events | within Day90

SECONDARY OUTCOMES:
Proportion of subjects with an excellent outcome defined by the functional assessments | Day 365
Proportion of subjects exhibiting functional outcome throughout the range of mRS scores by shift analysis | Day 90
Proportion of subjects exhibiting functional outcome throughout the range of mRS scores by shift analysis | Day 365
Proportion of subjects who meet all of a mRS score of ≤2, NIHSS score improvement of ≥75% from baseline and a BI score of ≥95 | Day 90
Proportion of subjects with a mRS score of ≤1 and a mRS score of ≤2 | Day 90
Proportion of subjects with a NIHSS score of ≤1 | Day 90
Proportion of subjects with a favorable outcome (NIHSS score improvement of ≥75% from baseline) in neurological symptoms | Day 90
Proportion of subjects with a BI score of ≥95 | Day 90
Proportion of subjects who survived without life-threatening adverse events (AEs) | Day 90
Proportion of subjects who survived without secondary infections | Day 90
Global recovery (i.e., GEE) and dichotomous assessment | Day 90
  Global recovery is an integrated assessment of patients who meet all of mRS score of ≤2, NIHSS score improvement of ≥75% from baseline, and BI score of ≥95, survival without life-threatening AEs and secondary infections
Comparison of the incidence of secondary infections (local and systemic), AEs, death, vital signs and laboratory parameters between the HLCM051 and the placebo groups | 1 year

OTHER OUTCOMES:
Changes in biomarkers (white blood cell populations and inflammatory markers) from baseline | Day 2, Day 7, Day 30.

CONTACTS AND LOCATIONS:
Locations (1):
- Hokkaido University Hospital, Sapporo, Japan

REFERENCES:
- [Derived] Houkin K, Osanai T, Uchiyama S, Minematsu K, Taguchi A, Maruichi K, Niiya Y, Asaoka K, Kuga Y, Takizawa K, Haraguchi K, Yoshimura S, Kimura K, Tokunaga K, Aoyama A, Ikawa F, Inenaga C, Abe T, Tominaga A, Takahashi S, Kudo K, Fujimura M, Sugiyama T, Ito M, Kawabori M, Hess DC, Savitz SI, Hirano T; TREASURE Study Investigators. Allogeneic Stem Cell Therapy for Acute Ischemic Stroke: The Phase 2/3 TREASURE Randomized Clinical Trial. JAMA Neurol. 2024 Feb 1;81(2):154-162. doi: 10.1001/jamaneurol.2023.5200. PMID 38227308
- [Derived] Osanai T, Houkin K, Uchiyama S, Minematsu K, Taguchi A, Terasaka S. Treatment evaluation of acute stroke for using in regenerative cell elements (TREASURE) trial: Rationale and design. Int J Stroke. 2018 Jun;13(4):444-448. doi: 10.1177/1747493017743057. Epub 2017 Nov 14. PMID 29134924